CLINICAL TRIAL: NCT07117006
Title: Anterior Open Bite Closure by Clear Aligners Versus Fixed Appliances in Adult Patients With Skeletal Open Bite: A Randomized Clinical Trial
Acronym: AOB-Mx_INT-MS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Shady Mohamed Ali Elkelany, Resident at International Orthodontic Program (IOP), Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CUFD-Ortho2025-001
Record Dates: First submitted 2025-08-05; First posted 2025-08-12 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Skeletal Open Bite; Open Bite; Maxillary Intrusion; Mini-screws; Clear Aligner Appliance
Keywords: Openbite; Skeletal anchorage; Fixed appliance; Aligners; Intrusion
MeSH Terms: conditions — Open Bite

STUDY DESIGN:
Masking Description: statistician will be blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- comparator- fixed appliance (Active Comparator): miniscrew-supported maxillary posterior segments' intrusion will be done using fixed appliances
  Interventions: Device: miniscrew- supported maxillary posterior segments' intrusion using clear aligners

INTERVENTIONS:
Device: miniscrew- supported maxillary posterior segments' intrusion using clear aligners — maxillary posterior segments will be intruded with the aid of miniscrews and clear aligners

SUMMARY:
Here's a 1,000-word (quarter-length) concise version of your research brief, preserving the key structure and essential details:

Brief Summary: Comparative Management of Skeletal Anterior Open Bite Using Mini-Screw Supported Intrusion with Clear Aligners Versus Fixed Appliances

PICO elements

Population: Adults (17-25 years) with uncompensated skeletal anterior open bite.

Intervention: TAD-supported intrusion with clear aligners. Comparison: TAD-supported intrusion with fixed appliances.

Outcomes:

Primary: Anterior open bite closure. Secondary: Molar intrusion, mandibular autorotation, incisor movement and quality of life.

DETAILED DESCRIPTION:
The aim of the study is to compare the effects of mini-screw supported maxillary posterior segments' intrusion using fixed appliances versus clear aligners.

ELIGIBILITY:
Inclusion Criteria:

* uncompensated skeletal openbite with normal incisal show at rest and smiling
* good oral hygeine

Exclusion Criteria:

* systemic disease
* extraction or missing dentition
* root resorption in posterior teeth
* carious or fractured upper posterior teeth peridontal affected upper posterior teeth

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2024-12-30 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Anterior open bite closure | 6 months
  the anterior open bite will be measured between the incisors using a digital caliper

SECONDARY OUTCOMES:
amount of maxillary posterior teeth intrusion | 6 months
  the distance between the molar tri-furcation/premolar center to the Frankfurt Horizontal plane
Amount of mandibular posterior teeth extrusion | 6 months
  the distance between molar bi-furcation or premolar center to the mandibular plane

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of dentistry, cairo university, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No